CLINICAL TRIAL: NCT06984419
Title: A Post-marketing, Open-label, Non-comparative, Multi-center Investigation to Evaluate the Effectiveness and Safety of a Medical Device "Alexa Volume" (DIACO BIOFARMACEUTICI S.r.l., Italy) Based on Cross-linked Hyaluronic Acid for Correction of the Midface Volume Los
Brief Title: Clinical Investigation of the Medical Device "Alexa Volume" for Correction of Midface Volume Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Hyalual GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D/Alexa.Vol.-2021
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Aesthetic; Aesthetic Rejuvenation; Midface Volumization; Age-related Volume Deficit in the Mid-face
Keywords: Age-related; midface; volume; facial aesthetic; Alexa Volume

STUDY DESIGN:
Intervention Model Description: This was a non-comparative, open-label study where all subjects received subcutaneous or upper-periosteal injections of Alexa Volume according to standardized procedures under routine clinical (cosmetology) conditions. No control or placebo group was included, and all participants were followed over 180 days for aesthetic and safety outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alexa Volume Treatment Arm (Experimental): Participants in this single treatment arm received subcutaneous or upper-periosteal injections of Alexa Volume, a CE-marked cross-linked hyaluronic acid gel, for the correction of midface volume loss. The initial injection was administered at Visit 1, with an optional additional correction at Visit 2 based on the Investigator's assessment. Effectiveness and safety evaluations were conducted through Visit 4 (Day 180).
  Interventions: Device: Cross-linked hyaluronic acid dermal filler

INTERVENTIONS:
Device: Cross-linked hyaluronic acid dermal filler — Alexa Volume is a CE-marked, cross-linked hyaluronic acid dermal filler used for aesthetic correction of midface volume loss. It was administered subcutaneously or to the upper periosteum in adult female participants according to standardized procedures.

SUMMARY:
This is a post-marketing, open-label, non-comparative, multi-center clinical investigation to evaluate the effectiveness and safety of the medical device "Alexa Volume" (DIACO BIOFARMACEUTICI S.r.l., Italy), based on cross-linked hyaluronic acid, for the correction of midface volume loss. The study involved 68 female subjects across Poland and Ukraine who received Alexa Volume injections in the midface area. Effectiveness was assessed using the Global Aesthetic Improvement Scale (GAIS), Wrinkle Severity Rating Scale (WSRS), and Medicis Midface Volume Scale (MMVS). The study demonstrated statistically significant improvements in aesthetic outcomes and confirmed a favorable safety profile with minimal adverse events

DETAILED DESCRIPTION:
This clinical investigation evaluated the effectiveness and safety of the CE-marked medical device "Alexa Volume," a cross-linked hyaluronic acid filler, for correction of midface volume loss in adult subjects. Conducted at multiple centers in Poland and Ukraine, the open-label, non-comparative study collected post-marketing data under routine clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Twenty-five (25) years of age or older at time of consent.
* Desire and willingness for correction or enhancement of his/her mid-face area.
* Subjects presenting with loss of volume and contour of the midface area 2 or more score according to MMVS bilaterally.
* Nasolabial folds severity grade 2 or more according to WSRS bilaterally.
* Treatment-naive subjects for fillers in the areas to be treated in the last 12 months, otherwise as decided by the Investigator.
* Subjects with signed informed consent and photo consent.
* Medical history and physical examination which, based on the Investigator's opinion, do not prevent the subject from taking part in the investigation and use the investigational medical device (IMD).
* Subjects not pregnant, non-breastfeeding.
* Subject must be willing to complete the entire course of the investigation.

Exclusion Criteria:

* Pregnant, planning pregnancy during the investigation or breastfeeding women.
* Subjects with known hypersensitivity to any compound of the IMD.
* Subjects with history of any other adverse effect, which could prevent the subject from participating in the investigation according to the Investigator's opinion.
* Any prior surgery, any prior cosmetic procedures or side effects from previous procedures in the injected area, including permanent fillers, that may interfere with the results.
* Subjects with presence of autoimmune disease or other chronic disease that in the opinion of the Investigator may interfere with the outcome of the investigation.
* Subjects with active inflammation or infection in the areas of Alexa administration.
* Subjects with tattoo and/or scar in the area of Alexa Volume administration that in the Investigator's opinion would interfere with investigation assessments.
* Subjects who tend to develop hypertrophic scarring.
* Subjects with impaired hemostatic function, which could prevent the subject from participating in the investigation according to the Investigator's opinion.
* Subjects with fibrosis, birthmark, or residual material in the area of intended use of Alexa Volume.
* Subjects participating in other clinical investigations within 30 days prior to the Visit 1.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Investigator-evaluated change in midface volume using the Global Aesthetic Improvement Scale (GAIS) from baseline (Visit 1) to Day 28 (Visit 3). | 28 days (from baseline Visit 1 to Visit 3)
  The GAIS (Global Aesthetic Improvement Scale) is a 5-point ordinal scale used to assess improvement in facial aesthetics. The scale ranges from 1 (Very Much Improved) to 5 (Worse), where lower scores indicate better outcomes. Investigators evaluated standardized photographs taken before and after treatment. A reduction of ≥1 point from baseline was considered a clinically meaningful improvement.

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (3):
  - Silmedic Sp. z o.o., Katowice
  - Provita Sp. z o.o., Katowice
  - Ośrodek Medyczny Osteomed s.c., Krakow
- Institute Hyalual LLC, Kyiv, Ukraine